CLINICAL TRIAL: NCT07334587
Title: Comparison of Efficacy and Safety Between FOLFOX-6 and CAPOX in Metastatic Colorectal Carcinoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Allama Iqbal Medical College (Other)
Responsible Party: Principal Investigator, Parnia Ansari, Principal Investigator, Allama Iqbal Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AllamaIqbalMC1
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Carcinoma (mCRC)
Keywords: Oxaliplatin; Metastatic colorectal cancer; Fluorouracil; Antineoplastic combined chemotherapy; Capecitabine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Platinum Compounds; Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CAPOX (Experimental): Participants will receive combination chemotherapy with capecitabine and oxaliplatin following standard dosing schedule after surgical management of metastatic colorectal carcinoma.
  Interventions: Drug: Capecitabine and Oxaliplatin
- Group FOLFOX-6 (Active Comparator): Participants will receive combination chemotherapy with fluorouracil, leucovorin calcium, and oxaliplatin following standard FOLFOX-6 protocol after surgical management of metastatic colorectal carcinoma.
  Interventions: Drug: Fluorouracil, Leucovorin Calcium, and Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine and Oxaliplatin — Oxaliplatin 130 mg per square meter administered intravenously on Day 1, together with oral capecitabine 1000 mg per square meter every 12 hours from Day 1 to Day 14.
  The treatment cycle will be repeated every 21 days for 6 to 8 cycles.
  Other Names: Fluoropyrimidine-based chemotherapy with platinum compound
  Arms: Group CAPOX
Drug: Fluorouracil, Leucovorin Calcium, and Oxaliplatin — Oxaliplatin 85 mg per square meter administered intravenously, leucovorin calcium 400 mg per square meter intravenous infusion, followed by fluorouracil bolus and continuous fluorouracil infusion over 46 hours at a dose of 2400 mg per square meter.
  The regimen will be repeated every 14 days for 12 cycles.
  Other Names: Oxaliplatin-based infusional fluoropyrimidine chemotherapy regimen
  Arms: Group FOLFOX-6

SUMMARY:
This randomized controlled trial is designed to compare the efficacy and safety of two commonly used chemotherapy regimens, FOLFOX-6 and CAPOX, in adults with metastatic colorectal carcinoma who are receiving chemotherapy after surgery at the Department of Oncology, Jinnah Hospital, Lahore. A total of 248 eligible patients aged 20 to 70 years will be enrolled using consecutive sampling and randomly allocated in equal numbers to receive either CAPOX or FOLFOX-6 according to standard dosing schedules. Participants will be followed for 3 months to determine whether meaningful differences exist between the two regimens in clinically important outcomes. The primary comparison will focus on disease progression within the follow-up period. Additional safety and treatment feasibility outcomes will include the need for chemotherapy dose reduction due to toxicity, treatment discontinuation, hepatotoxicity based on liver function abnormalities, diarrhea persisting for more than 3 days, and mortality during follow-up. The study hypothesis is that the outcomes of FOLFOX-6 and CAPOX differ in terms of effectiveness and adverse effects. The findings are expected to inform selection of a regimen that provides better disease control with fewer treatment-limiting side effects in the local clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-70 years,
* Both genders,
* Diagnosed with metastatic colorectal carcinoma, receiving chemotherapy after surgery.

Exclusion Criteria:

* Patients with non-metastatic disease at the time of diagnosis, coexisting other malignancy, and administration of adjuvant chemotherapy in an external center
* Patients with a history of neurologic disease (as per medical record)
* Patients already taking trial treatment or enrolled in another trial

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Disease progression | Within 3 months after initiation of assigned chemotherapy regimen
  Disease progression will be defined as an increase in lesion size and/or development of new symptoms consistent with worsening metastatic colorectal carcinoma, assessed clinically and by available follow-up evaluation during the follow-up period, as per the study operational definition.

SECONDARY OUTCOMES:
Hepatotoxicity | ithin 3 months after initiation of assigned chemotherapy regimen
  Hepatotoxicity will be defined as alanine aminotransferase and aspartate aminotransferase levels greater than two times the upper limit of normal and/or total bilirubin level greater than 5 milli-international units, occurring during follow-up, as per operational definition.
Diarrhea | Within 3 months after initiation of assigned chemotherapy regimen
  Diarrhea will be defined as loose, watery stools persisting for more than 3 days during the follow-up period.
Discontinuation of chemotherapy | Within 3 months after initiation of assigned chemotherapy regimen
  Permanent stopping of the assigned chemotherapy regimen due to severe adverse effects during the follow-up period.
All-cause mortality | Within 3 months after initiation of assigned chemotherapy regimen
  Death from any cause occurring during the 3-month follow-up period after initiation of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Parnia Ansari, Principal Investigator — Allama Iqbal Medical College, Lahore
Locations (1):
- Allama Iqbal Medical College, Lahore, Lahore, Punjab Province, Pakistan